CLINICAL TRIAL: NCT01222754
Title: A Phase I Trial of Lenalidomide and Radiotherapy in Children With Diffuse Intrinsic Pontine Gliomas and High-grade Gliomas
Brief Title: Lenalidomide and Radiation Therapy in High Grade Gliomas or Diffuse Intrinsic Pontine Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100219; 10-C-0219; NCT01226940 (obsolete NCT alias)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Anaplastic Astrocytoma; High Grade Glioma
Keywords: Newly Diagnosed; DIPG; Radiation Therapy; CC-5013; XRT; Brain Tumor; Glioma; Pediatrics
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Astrocytoma; Glioma; Brain Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Radiation with Lenalidomide
  Interventions: Drug: Lenalidomide; Radiation: XRT, 54-59.4 Gy

INTERVENTIONS:
Drug: Lenalidomide — 1. With radiation therapy five days per week, concurrent doses of lenalidomide daily in a standard Phase I dose escalation design.
  2. Maintenance dosing of lenalidomide, post-radiation, for 21 days of a 28 day course.
Radiation: XRT, 54-59.4 Gy — Radiation therapy five days per week to a prescription dose of 54-59.4 Gy, with concurrent administration of lenalidomide

SUMMARY:
Background:

- Children who are diagnosed with brain tumors known as high grade gliomas or diffuse intrinsic pontine gliomas are generally treated with radiation therapy and chemotherapy. However, these tumors are very difficult to cure, and the tumor frequently begins to grow again even after treatment or surgery. Researchers are interested in determining whether the anticancer drug lenalidomide, which has been used to treat other aggressive types of cancer, is a safe and effective additional treatment for children who are scheduled to receive radiation therapy to treat high grade gliomas or diffuse intrinsic pontine gliomas.

Objectives:

- To determine the safety and effectiveness of lenalidomide, in conjunction with radiation therapy, as a treatment for children who have been diagnosed with high grade gliomas or diffuse intrinsic pontine gliomas.

Eligibility:

- Children and adolescents up to 21 years of age who have been diagnosed with high grade gliomas or diffuse intrinsic pontine gliomas and have not had radiotherapy or chemotherapy.

Design:

* Participants will be screened with a medical history, physical examination, blood and urine tests, and imaging studies.
* Participants will have two phases of treatment: a lenalidomide plus radiation phase and a lenalidomide-only phase.
* During the radiation phase, participants will take lenalidomide daily and have 6 weeks of radiation therapy (five treatments per week). After the radiation therapy, participants will stop taking lenalidomide for 2 weeks before continuing to the next phase.
* During the lenalidomide-only phase, participants will take lenalidomide daily for 21 days, followed by 7 days without lenalidomide (28-day cycle of treatment). Participants will have up to 24 cycles of lenalidomide.
* Participants will have frequent blood tests during the first cycle of treatment, and will have imaging studies or other tests as required by the study researchers.
* Treatment will continue until the disease progresses, the participant chooses to leave the study, or the researchers end the study.

DETAILED DESCRIPTION:
Background:

Brain tumors are the most common solid neoplasm in childhood and the second most common group of pediatric cancers.

Standard therapeutic options for brain tumors consist of surgical resection, radiation therapy and chemotherapy; yet overall survival rates for malignant brain tumors remain low.

Radiation therapy plays a key role in the treatment of diffuse intrinsic pontine gliomas (DIPG) and high-grade gliomas (HGG), and thalidomide has been shown in an animal model to be a radiosensitizer.

Lenalidomide, a thalidomide analog with antiangiogenic, cytotoxic and immunomodulatory effects, is being evaluated for the treatment of CNS tumors, and has shown tolerability and activity in pediatric studies.

Objectives:

To determine the tolerability and toxicity profile of oral lenalidomide when administered to children with newly diagnosed HGG and DIPG with concurrent radiation at doses up to 116 mg/m(2)/day.

To evaluate long-term tolerability of lenalidomide in children with newly-diagnosed HGG and DIPG.

To evaluate magnetic resonance imaging (MRI) sequences for noninvasive monitoring of metabolic and biologic changes in malignant brain tumors with therapy.

To estimate 6 month and 12 month progression free survival (PFS) and overall survival (OS) in this patient population.

To determine if angiogenic and/or immunomodulatory biomarkers in the blood and urine correlate with toxicity and disease response.

To determine the rate of CNS metastatic disease in patients treated with antiangiogenic chemotherapy.

To determine any correlation of steady state pharmacokinetics of lenalidomide with time to progression, number and type of toxicities, and dose limiting toxicities.

Eligibility:

Children with newly diagnosed HGG or DIPG, less than 22 years of age, no prior chemotherapy or radiation therapy, and performance score greater than or equal to 60%.

Children with HGG must have an inoperable or incompletely resected tumor.

Clinical laboratory tests must be within stated limits.

Design:

There will be two phases to therapy on this study, the Radiation Phase and the Maintenance Phase. The MTD will be determined by tolerability during the Radiation Phase.

Eligible patients will receive radiation therapy five days per week to a prescription dose of 54-59.4 Gy, with concurrent administration of lenalidomide daily in a standard Phase I dose escalation design.

At the conclusion of radiation therapy, there will be a two week break followed by maintenance dosing of lenalidomide for 21 days of a 28 day course, until unacceptable toxicity, disease progression or completion of 24 courses of lenalidomide beyond radiotherapy (unless otherwise approved by PI).

Using a multi-center, standard phase I dose escalation design, the total sample size

and the study duration are expected to be 18 - 30 patients and 5-6 years, respectively.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Histological diagnosis:

* Histological confirmation of a high-grade malignant glioma is required. Histologic diagnoses include, but are not limited to, anaplastic astrocytoma and glioblastoma multiforme. Patients with DIPG are exempt from histologic verification if they have typical MRI findings of DIPG (i.e. hypo- or isointense on T1-weighted imaging, hyperintense on FLAIR or T2-weighted imaging, epicenter in the pons, greater than 50% of pons involved) in the face of a typical clinical presentation.
* Inoperable tumor or residual disease after resection

Prior therapy:

-No prior chemotherapy or radiation therapy for HGG or DIPG is permitted. Prior chemotherapy or radiation therapy for treatment of other malignancies is permitted.

Age:

-Patients must be less than 22 years of age at the time of diagnosis.

Able to swallow capsules whole

Performance Score:

-Patients should have a Karnofsky/Lansky score of greater than or equal to 60. Patients who require special assistance due to tumor-related paralysis, but who are out of bed during the day will be considered ambulatory for the purpose of calculating the performance score. Patients must be able to communicate any symptoms.

Laboratory Evaluation:

* The following laboratory values must be assessed within seven (7) days prior to the start of therapy. Laboratory tests should be repeated within 48 hours of beginning therapy if there has been a significant clinical change.
* Patients must have adequate organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than 1.5 times upper limit of normal
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * creatinine below age-adjusted maximum limits below

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m(2)
* Age (Years) Maximum Serum Creatinine (mg/dl):

  * Less than or equal to 5 years; 0.8
  * Age greater than 5, but less than or equal to 10 ; 1.0
  * Age greater than 1, but less than or equal to 15 ; 1.2
  * Less than 15 years of age; 1.5

Females only:

* urine or serum pregnancy test negative
* No overt renal, hepatic, cardiac or pulmonary disease.

Steroids:

-Newly diagnosed patients may need to be on steroids due to surgery or control of neurologic symptoms. Patients on steroids postoperatively or for control of tumor-related edema are eligible, but attempts to keep patients on the lowest dose necessary to control symptoms should be made.

Patients of childbearing potential:

-Female Subjects:

* Definition of female of childbearing potential (FCBP)

This protocol defines a female of childbearing potential as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

--Criteria for female children of childbearing potential (FCCBP)

This protocol defines FCCBP as females who have:

* Achieved menarche and/or breast development in Tanner stage 2 or greater

  ----Onset of fertility typically occurs within 3-12 months after menarche. Menarche varies considerably from person to person, and thus no age cut off can be attributed. One of the primary tools used to follow a girl s progress through puberty is the Tanner staging system, which describes the pattern of development of the secondary sex characteristics. Tanner stage 2 corresponds to the beginning of breast development, which is the first visible sign of puberty in girls. Breast development is estrogen stimulated, and since ovulation cannot occur without estrogen, Tanner stage 2 will be a reliable marker for the definition of fertility.
* Has not undergone a hysterectomy or bilateral oophorectomy.

Note: Amenorrhea following cancer therapy does not rule out childbearing potential

--Criteria for female children not of childbearing potential (FCNCBP)

This protocol defines FCNCBP as females:

* Who have not yet experienced menarche or breast development in Tanner stage 2.
* Who have undergone a hysterectomy or bilateral oophorectomy.

Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 14 days and again within 24 hours prior to starting Course 1 of lenalidomide. Further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy. A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). All patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure.

-Male Subjects:

* Appropriate male subjects (i.e. those who have reached puberty and are sexually active) will be counseled regarding birth control methods. They must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
* Appropriate male patients will be given a reproductive risks handout and counseled by a provider. For sexually active patients, the counseling session, consent and counseling checklist will be documented monthly.

Informed consent:

All patients or their legal guardians (if the patient is less than18 years old) or durable power of attorney (DPA) must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study. When appropriate, pediatric patients will be included in all discussions in order to obtain verbal assent.

In the event that the patient and/or the patient s parents are unable to travel to NIH should re-consenting be necessary, a telephone consent may be performed by the principal investigator according to Clinical Center Policy M77-2. The telephone consent will be

witnessed by a member of the research team who is on the telephone with the patient and PI and who can confirm the patient s consent to participate. A copy of the signed consent will be mailed to the participant. The consenting process will be documented in the

patient s record which is signed by the PI and co-signed by the witness to the consent.

Durable Power of Attorney:

Assignment of DPA to a family member or guardian should be offered to all patients 18 years of age.

Signed informed consent according to institutional guidelines must be obtained.

EXCLUSION CRITERIA:

Patients who have had prior chemotherapy for this tumor.

Patients with an HGG that was completed resected with good margins.

Patients with a body surface area (BSA) less than or equal to 0.4 m(2) are excluded because the lowest dose of the medication is 5 mg in capsule form.

Patients with a known coagulation disorder are excluded. Patients with a first-degree relative with a history of venous thrombosis before age 50 yrs or an arterial thrombosis before age 40 yrs must have the following testing performed prior to enrollment to exclude a heritable disorder. Patients with a suspected disorder will be excluded due to the potential increased risk of thrombosis.

Patients who have had a thromboembolic event that is not line-related are excluded.

Patients with any significant medical illnesses that, in the investigator s opinion, cannot be adequately controlled with appropriate therapy, would compromise a patient s ability to tolerate this therapy or result in inability to assess toxicity. This includes, but is not limited to uncontrolled intercurrent illness including ongoing or active infection, cardiac disease, renal impairment or psychiatric illness/social situations that would limit compliance with study requirements.

Patients with a history of Toxic Epidermal Necrolysis (TEN) or Stevens-Johnson syndrome are excluded as this has occurred in patients receiving lenalidomide.

Patients receiving any other investigational agents.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide (i.e. thalidomide).

Patients with known hypersensitivity to anhydrous lactose, microcrystalline cellulose, croscarmellose sodium, and magnesium stearate.

Pregnant or breast feeding females:

Pregnant women are excluded from this study because lenalidomide is in a class with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide.

Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lenalidomide. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Patients identified as needing spinal radiation at diagnosis (e.g. spinal metastasis or malignant cells identified on CSF cytology) are excluded due to the increased risk of myelosuppression.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2010-11-23 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Tolerability | 2 years
  The plasma steady state concentration (and CSF levels if available for other reasons) will be correlated with toxicities (type and incidence), time to progression and response.
Toxicity Profile | 2 years
  We will also estimate the population parameters using nonlinear mixed effects modeling methods (NONMEM)

SECONDARY OUTCOMES:
Evaluate MRI Sequences | 3 years
Progression-free survival | 4 years
Overall Survival | 4 years
Biomarkers & toxicity/disease response correlation | 3 years
Pharmacokinetics correlation with progression and toxicities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John W Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Siffert J, Greenleaf M, Mannis R, Allen J. Pediatric brain tumors. Child Adolesc Psychiatr Clin N Am. 1999 Oct;8(4):879-903, x. PMID 10553209
- [Background] Finlay JL, Boyett JM, Yates AJ, Wisoff JH, Milstein JM, Geyer JR, Bertolone SJ, McGuire P, Cherlow JM, Tefft M, et al. Randomized phase III trial in childhood high-grade astrocytoma comparing vincristine, lomustine, and prednisone with the eight-drugs-in-1-day regimen. Childrens Cancer Group. J Clin Oncol. 1995 Jan;13(1):112-23. doi: 10.1200/JCO.1995.13.1.112. PMID 7799011
- [Background] Freeman CR, Farmer JP. Pediatric brain stem gliomas: a review. Int J Radiat Oncol Biol Phys. 1998 Jan 15;40(2):265-71. doi: 10.1016/s0360-3016(97)00572-5. PMID 9457808
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0219.html